CLINICAL TRIAL: NCT04671251
Title: A Multicenter, Open-Label, Dose-Escalation Phase 1b Study of AEVI-007 in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Phase 1b Study of AEVI-007 in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AEVI-007-MM-101
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AEVI-007 (Experimental): Open-label, dose-escalation, single-arm
  Interventions: Drug: AEVI-007

INTERVENTIONS:
Drug: AEVI-007 — 50 mg of AEVI-007 and will be reconstituted with 1.2 mL of water for injection.

SUMMARY:
This is a multicenter, open-label, dose-escalation Phase 1b study of AEVI-007 in subjects with relapsed or refractory Multiple Myeloma.

The objectives of the study are to evaluate the safety, pharmacokinetics and pharmacodynamics of AEVI-007.

DETAILED DESCRIPTION:
This was a multicenter, open-label, dose-escalation, sequential groups Phase 1b clinical study in subjects with R/R multiple myeloma. The study utilized a "3+3" design. Three subjects were enrolled at each dose, starting with the initial dose of 4 mg/kg. If there were no DLTs, escalation to the next cohort took place. If there was 1 DLT, then the cohort was to be expanded to 6. If there were no further DLTs, then escalation to the next dose took place. If there were 2 DLTs in the initial 3 subjects, or 2 in the expanded cohort of 6 subjects, then the maximally tolerated dose (MTD) had been exceeded and dose escalation stopped. The dose prior to the dose where DLT was observed was then the RP2D. To allow safety assessment, the dosing of subjects within each dose level was staggered, with at least 24 hours between each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has active R/R multiple myeloma.
2. Subject has measurable myeloma based on any of the following:

   * Serum M-protein > 0.5 g/dL
   * Urine M-protein > 200 mg/24 hours
   * Serum free light chains > 10 mg/dL
   * Measurable plasmacytoma or extramedullary disease
3. Subject has active myeloma despite prior therapy with a proteasome inhibitor, an immunomodulatory agent and an anti-CD38 antibody.

   Note: Subject must not be a candidate for regimens known to provide clinical benefit.
4. Subject has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
5. Subject is > 18 years of age.
6. Subject has adequate hematopoietic, renal and hepatic function, defined as:

   * Absolute neutrophil count > 1,000/μL; platelet count > 75,000/μL in patients with < 50% marrow involvement
   * Absolute neutrophil count > 750/μL; platelet count > 50,000/μL in patients with >50% marrow involvement
   * Serum creatinine < 2.5 mg/dL or calculated creatinine clearance of > 30 mL/min according to the Cockcroft-Gault equation
   * Aspartate transaminase/alanine transaminase ≤2.5× the upper limit of normal (ULN) and total bilirubin < 2× the ULN
7. If applicable, the subject has undergone prior autologous hematopoietic stem cell transplantation more than 100 days prior to the Screening Visit.
8. Female patients of childbearing potential who are heterosexually active and male patients with female sexual partners of childbearing potential must agree to use an effective method of contraception (eg, oral contraceptives, double-barrier methods such as a condom and a diaphragm, intrauterine device) or abstain from sexual activity during the study and for 220 days (5 half-lives) following the last dose of study medication, or to abstain from sexual intercourse for this duration of study participation. A woman not of childbearing potential is one who has undergone bilateral oophorectomies or who is post-menopausal, defined as the absence of menstrual periods for 12 consecutive months.
9. Subject has provided written informed consent for this study.

Exclusion Criteria:

1. Subject has currently active infection requiring use of systemic antimicrobial therapy.
2. Subject has received corticosteroids (>10 mg/daily prednisone or equivalent) or chemotherapy within 2 weeks of study drugs (4 weeks for nitrosourea, melphalan or monoclonal antibodies).
3. Subject has hyperviscosity syndrome.
4. Subject has central nervous system involvement by myeloma, including leptomeningeal involvement.
5. Subject is judged to be at risk for impending fracture.
6. Subject has known amyloidosis or POEMS (Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, Skin changes) syndrome.
7. Subject had another malignancy within 1 year of study entry with high probability of recurrence.
8. Subject is pregnant or lactating.
9. Subject has a history of, or tests positive for, hepatitis B, untreated hepatitis C or human immunodeficiency virus (HIV). Subject with hepatitis C who has received a full course of anti-viral therapy or who is currently receiving anti-viral therapy with undetectable levels of hepatitis C RNA is eligible for the trial.
10. Subject has undergone major surgery or trauma within 4 weeks of study entry.
11. Subject has been previously treated with an anti IL 18 antibody.
12. Subject is currently taking immunomodulatory drugs, including pharmacologic doses of systemic glucocorticoids (> 10 mg prednisone daily or equivalent), anti tumor necrosis factor alpha (TNFα) antibodies, anti-IL-17 antibodies, anti IL 12/23 antibodies, phosphodiesterase-4 (PDE-4) inhibitors, janus kinase (JAK) inhibitors, IL-6 inhibitors, rituximab, methotrexate, cyclosporine, mycophenolate.
13. Subject with known active autoimmune disorders including, but not limited to, rheumatoid arthritis, lupus, systemic sclerosis, Sjogren's syndrome, psoriatic arthritis, ulcerative colitis, Crohn's disease, vasculitis, multiple sclerosis. Subjects with autoimmune endocrinopathies on stable doses of replacement hormone therapy are eligible for the trial.
14. Subject has had a prior allogeneic transplant.
15. Subject has New York Heart Association (NYHA) Class III or IV Congestive Heart Failure (CHF), myocardial infarction or acute coronary syndrome within 6 months prior to the Screening Visit, ongoing angina pectoris, severe peripheral vascular disease, or any other concomitant medical disorder that might interfere with the subject's participation in the trial or interpretation of the study data.
16. Subject has psychiatric, substance abuse or social conditions that would interfere with the subject's participation or cooperation with the requirements of the trial.
17. Subject has known hypersensitivity to any of the components of AEVI-007.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose | Cohorts 1-3 will take approximately 4-5 months
  Identify the recommended Phase 2 dose based on safety, pharmacokinetics and pharmacodynamics observed in this Phase 1b study.

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Approximately 9 months
Incidence of Clinically Significant Changes in Clinical Laboratory Results | Approximately 9 months
Incidence of Clinically Significant Changes in Vital Signs | Approximately 9 months
Incidence of Clinically Significant Changes in Electrocardiogram Recordings | Approximately 9 months
Incidence of Clinically Significant Changes to Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score | Approximately 9 months
Incidence of Clinically Significant Changes in Physical Examination Findings | Approximately 9 months
Maximum Observed Concentration of AEVI-007 | Approximately 9 months
Apparent Terminal Half-Life of AEVI-007 | Approximately 9 months
Clearance of AEVI-007 | Approximately 9 months
Volume of Distribution of AEVI-007 | Approximately 9 months
Area Under the Concentration-Time Curve From Time 0 to Time t of AEVI-007 | Approximately 9 months
Anti-myeloma activity | Approximately 9 months
  To assess the anti-myeloma activity of AEVI-007 based on International Myeloma Working Group (IMWG) criteria for response
Determination of ADAs | Approximately 9 months
  To determine the incidence of anti-drug antibodies to AEVI-007.
Time to Response (TTR) | Approximately 9 months
  Defined as the time from start of the treatment to the first observation of PR or better. TTR is restricted to only subjects with confirmed responses.
Progression Free Survival (PFS) | Approximately 9 months
  Defined as the duration from start of the treatment to disease progression or death (regardless of cause of death), whichever comes first
Duration of Response | Approximately 9 months
  Defined as the duration from the first observation of PR to the time of disease progression, with deaths from causes other than progression censored

CONTACTS AND LOCATIONS:
Overall Officials: Manish Patel, MD, Principal Investigator — Florida Cancer Specialist
Locations (7):
- United States (7):
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - James R. Berenson, MD., Inc., West Hollywood, California
  - Florida Cancer Specialists, Lake Mary, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Levine Cancer Institute, Charlotte, North Carolina
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No